CLINICAL TRIAL: NCT07298369
Title: Cracking Consciousness Study With Monroe & Neuphoria (Cohort 2&3)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 45835
Record Dates: First submitted 2025-12-05; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single arm where participants act as their own control
  Interventions: Device: Neuphoria Wearable

INTERVENTIONS:
Device: Neuphoria Wearable — Neuphoria wearable measures Electroencephalography (EEG) brainwaves.

SUMMARY:
In partnership with Monroe, this EEG neurofeedback study is looking at the efficacy of Neuphoria with Monroe for mental clarity and well-being.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to explore the efficacy of the Neuphoria neurofeedback device in enhancing cognitive performance and achieving peak mental states through advanced EEG technology. By monitoring brainwave activity in real-time, this trial aims to provide personalized feedback to participants, enabling them to train their brains for improved focus, creativity, and flow states. The device serves as a comprehensive brain optimization platform, offering personalized assessments, data-driven insights, and actionable recommendations for mental well-being.

In an era where mindfulness and meditation are highly valued, yet rarely quantified, this study collaborates with Neuphoria to venture into measuring higher states of consciousness, blending scientific rigor with the art of introspection. The objective is to transform beliefs and anecdotal evidence about consciousness and mental wellness into empirical data, thereby redefining our understanding of mental health.

Participants in this study are guided through an exploration of their mental landscapes, with the goal of capturing data that reflects their journey towards higher consciousness. Through engagement with meditation and mindfulness techniques, participants will be able to gain insights into their stress levels and mindfulness tendencies. These insights will be quantified through established tools such as the Perceived Stress Scale and the Freiburg Mindfulness Inventory, offering a structured pathway to personal mental wellness enhancement and elevated consciousness.

The primary aim of this trial is to objectively measure shifts in consciousness in participants using EEG data, in conjunction with traditional mindfulness and stress metrics. By providing personalized insights into how meditation and mindfulness practices affect mental health, the study empowers participants to make informed decisions about their self-care routines and investments in personal development.

The significance of this study lies in its potential to convert subjective experiences of meditation into objective, quantifiable data. This endeavor bridges the gap between belief and measurable outcomes, advancing our understanding of how mindfulness practices influence consciousness and mental health. While acknowledging the limitations in the universal applicability of the results, the personalized insights gleaned from this study promise to be invaluable for participants eager to deepen their mindfulness practice and achieve a state of equanimity. Through this remotely conducted trial, we aim not only to explore the boundaries of mental wellness but also to offer a scientifically grounded pathway for individuals seeking to optimize their mental states.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

* Individuals with severe mental health disorders
* Individuals with low frustration tolerance
* Individuals without access to emergency medical care
* Individuals involved in regulated professions
* Individuals with skepticism towards digital monitoring
* Individuals without a support system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
EEG Spectral Power by Frequency Band | Change from baseline (Day 1-7) in cognitive profile metrics at 4 to 5 weeks after the start of the intervention
  Electroencephalography (EEG) will be used to quantify spectral power across standard frequency bands (delta [1-4 Hz], theta [4-8 Hz], alpha [8-12 Hz], beta [12-30 Hz]). Power values will be derived using proprietary signal processing algorithms and summarized as relative power per band.
Perceived Stress Scale (Past Week Version) | Change from baseline (Day 1-3) in perceived stress levels at 4 to 5 weeks after the start of the intervention
  The Perceived Stress Scale (Past Week Version) is a modified version of the classic stress assessment tool that evaluates stress levels based on recent experiences within the last week. This scale helps in understanding how various situations have recently affected an individual's feelings and perceived stress levels. By focusing on a shorter time frame, it provides a more immediate assessment of stress, which can be particularly useful for quickly evaluating the effectiveness of stress management strategies or interventions. The tool retains its original structure, ensuring its reliability while making it more relevant for current stress evaluation.
  Score Range
  Minimum: 0
  Maximum: 40
  Interpretation
  Higher scores indicate worse outcomes, reflecting greater perceived stress over the past week.
Freiburg Mindfulness Inventory | Change from baseline (Day 1-3) in mindfulness levels at 4 to 5 weeks after the start of the intervention
  The Freiburg Mindfulness Inventory (FMI) is a valid and reliable questionnaire designed to measure mindfulness. The 14 items in the inventory cover all aspects of mindfulness. Participants are asked to reflect on their experiences over a certain period of time and answer each statement as honestly and spontaneously as possible. There are no 'right' or 'wrong' answers, the focus is solely on personal experience.
  Score Range
  The range depends on the version used:
  14-item version (FMI-14):
  Minimum: 14
  Maximum: 56
  Interpretation
  Higher scores indicate better outcomes, reflecting greater levels of mindfulness.
  Lower scores indicate lower mindfulness.
EEG-Derived Cognitive State Index | Change from baseline (Day 1-7) in cognitive profile metrics at 4 to 5 weeks after the start of the intervention
  A composite cognitive state index derived from EEG spectral features, reflecting participant alertness and engagement. The index is calculated using a proprietary algorithm and reported on a normalized scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=45810